CLINICAL TRIAL: NCT00070707
Title: Efficacy and Safety of Nasonex vs. Placebo in Subjects With SAR and Concomitant Asthma
Brief Title: Nasonex Compared With Placebo in Participants With Seasonal Allergic Rhinitis (SAR) and Concomitant Asthma (P03280)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Integrated Therapeutics Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03280; MK-0887-064 (Other: Merck)
Record Dates: First submitted 2003-10-07; First posted 2003-10-10 (Estimated); Results first posted 2019-07-18 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal; Asthma
Keywords: Seasonal Allergic Rhinitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Asthma | interventions — Mometasone Furoate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mometasone (Experimental): Mometasone nasal spray 200 mcg, administered once daily (QD) for 4 weeks
  Interventions: Drug: Mometasone; Drug: Albuterol/Salbutamol
- Placebo (Placebo Comparator): Matching placebo nasal spray, administered QD for 4 weeks
  Interventions: Drug: Placebo; Drug: Albuterol/Salbutamol

INTERVENTIONS:
Drug: Mometasone — Mometasone nasal spray 200 mcg/day administered as 2 sprays (50 mcg/spray) in each nostril.
  Other Names: Nasonex
  Arms: Mometasone
Drug: Placebo — Matching placebo nasal spray, administered QD as 2 sprays in each nostril.
  Arms: Placebo
Drug: Albuterol/Salbutamol — Albuterol/salbutamol metered dose inhaler (90 mcg/puff) used as needed as asthma rescue medication.
  Other Names: Proventil HFA

SUMMARY:
This study will compare mometasone nasal spray to placebo in treating the nasal and asthma symptoms experienced by participants with seasonal allergic rhinitis (SAR) and concomitant asthma.

ELIGIBILITY:
Inclusion Criteria:

* Have at least a two-year history of seasonal allergic rhinitis and an increase in asthma symptoms associated with the allergy season under study
* Demonstrate an increase in absolute FEV 1 less than 12%, with an absolute volume increase of at least 200 ml, after reversibility testing within the past 12 months
* Is skin test positive (skin prick test with a wheal diameter at least 3 mm larger than the diluent control or intradermal testing with the wheal diameter at least 7 mm larger than diluent control) at screening, or within 12 months prior to the screening visit, to a seasonal allergen (which may include seasonal molds) prevalent during the study period.
* Female participants of childbearing potential use a medically accepted method of birth control and agree to continue its use during the study or be surgically sterilized (eg, hysterectomy or tubal ligation). Females who are not sexually active at time of study agree and consent to use a medically acceptable method of birth control should they become sexually active while participating in the study.

Exclusion Criteria:

* Female participants who are pregnant, intend to become pregnant during the duration of the study, or are nursing.
* Have asthma symptoms and require chronic use of inhaled or systemic corticosteroids.
* Have current or historical frequent (2 or more episodes per year for the past 2 years), clinically significant sinusitis or chronic purulent postnasal drip.
* Have recent nasal septum ulcers, nasal surgery or nasal trauma, which should not be included until healing occurs.
* Have rhinitis medicamentosa or chronic obstructive pulmonary disease (COPD).
* Have an upper or lower respiratory tract or sinus infection that requires antibiotic therapy, or have a viral upper or lower respiratory infection.
* Have nasal structural abnormalities, including large nasal polyps and marked septum deviation, that significantly interferes with nasal air flow.
* Are dependent on nasal topical antihistamines, or nasal steroids.
* On immunotherapy (desensitization therapy) and will receive an increase in dose during the study; participants who will receive desensitization treatment within 24 hours prior to a study visit.
* Is a participant who smokes, or is an ex-smoker who has smoked within the previous six months.
* Is an investigator, study staff member, or family member involved with this study.
* Has active or quiescent tuberculosis infection of the respiratory tract, untreated fungal, bacterial, or systemic viral infections, or herpes simplex.
* Is a participant whose ability to provide informed consent is compromised.
* Has a history of non-compliance with medications or treatment protocols.
* Is morbidly obese (BMI >35).
* Is a night-shift worker or does not have a standard asleep at night/awake during the day cycle.
* Has any history of life-threatening asthma attacks or is treated in the emergency room or admitted to the hospital for asthma control within the previous 3 months or more than once in the previous 6 months

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2003-04-03 (Actual); Primary Completion 2003-11-26 (Actual); Study Completion 2003-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medial Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mometasone | Placebo
Started | 113 | 75
Completed | 99 | 68
Not Completed | 14 | 7
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 4 | 1
Not completed — Protocol Violation | 8 | 4
Not completed — Unrelated to Study Medication | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant in the mometasone treatment group did not have any post-baseline assessment and was excluded from the Intent-to-Treat (ITT) population, for which baseline demograpic characteristics were summarized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone | Placebo | Total
Number analyzed (Participants) | 112 | 75 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (12.2) | 31.8 (10.9) | 32.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 55 | 132
  Male | 35 | 20 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 83 | 60 | 143
  Black or African American | 22 | 8 | 30
  Hispanic | 5 | 6 | 11
  Asian | 1 | 1 | 2
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning (AM) and Evening (PM) Total Asthma Symptom Severity (TASS)
Description: Each morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her asthma symptoms. The TASS was the sum of severity scores for 4 asthma symptoms: cough, wheeze, difficulty of breathing, and chest tightness. The severity of each asthma symptom was rated on a 4-point scale (0=no symptom; 3=severe); minimum TASS=0; maximum TASS=12. A decrease in TASS indicated an improvement in asthma symptoms. The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 6.5 (0.22) | 5.9 (0.26)
  Change at Week 1 (AM) | -0.9 (0.20) | -1.4 (0.23)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -1.5 (0.26) | -1.5 (0.30)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -2.4 (0.26) | -2.1 (0.29)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -2.5 (0.27) | -2.6 (0.31)
  Change at Final Week (AM) | -2.2 (0.25) | -2.2 (0.29)
  Baseline (PM) | 6.6 (0.22) | 6.0 (0.26)
  Change at Week 1 (PM) | -1.4 (0.19) | -1.7 (0.22)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -1.7 (0.24) | -1.7 (0.28)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -2.6 (0.24) | -2.3 (0.28)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -2.7 (0.27) | -2.5 (0.31)
  Change at Final Week (PM) | -2.4 (0.25) | -2.4 (0.29)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.101, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.168, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.930, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.487, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.914, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.977, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.109, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.291, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.984, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.373, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.623, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.978, ANOVA

2. Secondary Outcome: Change From Baseline in AM and PM Cough Symptom Score
Description: Cough is an asthma symptom assessed by participants who used diary cards to record morning and evening cough (recorded twice daily). Every morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her coughing for the time period since the last evaluation (or for the previous 12 hours for the first evaluation). Cough was rated on a 4-point scale (0=no symptoms [best score] to 3=symptoms were hard to tolerate and interfered with daily life activity [worst score]). Reduction in score indicated an improvement in cough symptoms. The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 1.7 (0.07) | 1.5 (0.08)
  Change at Week 1 (AM) | -0.3 (0.05) | -0.3 (0.06)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -0.4 (0.07) | -0.4 (0.08)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -0.7 (0.08) | -0.4 (0.09)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -0.7 (0.08) | -0.5 (0.10)
  Change at Final Week (AM) | -0.6 (0.08) | -0.5 (0.09)
  Baseline (PM) | 1.7 (0.07) | 1.5 (0.08)
  Change at Week 1 (PM) | -0.4 (0.06) | -0.4 (0.07)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -0.5 (0.07) | -0.4 (0.09)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -0.7 (0.08) | -0.5 (0.09)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -0.7 (0.09) | -0.6 (0.10)
  Change at Final Week (PM) | -0.6 (0.08) | -0.6 (0.09)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.023, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.693, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.483, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.088, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.210, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.178, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.055, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.915, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.471, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.110, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.305, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.461, ANOVA

3. Secondary Outcome: Change From Baseline in AM and PM Wheeze Symptom Score
Description: Wheezing is a symptom of asthma. The wheezing assessment was based on participant diary data only. Every morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her wheezing for the time period since the last evaluation (or for the previous 12 hours for the first evaluation). Wheeze severity was rated on a 4-point scale (0=no wheezing [best score] to 3=wheezing was hard to tolerate and interfered with daily life activity [worst score]). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 1.5 (0.07) | 1.3 (0.09)
  Change at Week 1 (AM) | -0.2 (0.05) | -0.3 (0.06)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -0.4 (0.08) | -0.3 (0.09)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -0.6 (0.08) | -0.5 (0.08)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -0.6 (0.08) | -0.6 (0.09)
  Change at Final Week (AM) | -0.5 (0.07) | -0.5 (0.09)
  Baseline (PM) | 1.5 (0.08) | 1.3 (0.09)
  Change at Week 1 (PM) | -0.3 (0.06) | -0.4 (0.07)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -0.4 (0.07) | -0.4 (0.08)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -0.6 (0.07) | -0.5 (0.08)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -0.7 (0.08) | -0.6 (0.09)
  Change at Final Week (PM) | -0.6 (0.07) | -0.5 (0.09)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.068, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.116, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.749, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.289, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.982, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.941, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.128, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.484, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.673, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.250, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.450, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.774, ANOVA

4. Secondary Outcome: Change From Baseline in AM and PM Difficulty Breathing Symptom Score
Description: Difficulty breathing is an asthma symptom assessed by participants using diary cards to record morning and evening difficulty breathing (recorded twice daily). Every morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her difficulty breathing for the time period since the last evaluation (or for the previous 12 hours for the first evaluation). Difficulty breathing was rated on a 4-point scale (0=no symptom [best score] to 3=symptoms were hard to tolerate and interfered with daily life activity [worst score]). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 1.7 (0.06) | 1.6 (0.07)
  Change at Week 1 (AM) | -0.3 (0.06) | -0.3 (0.07)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -0.4 (0.07) | -0.4 (0.08)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -0.7 (0.07) | -0.6 (0.08)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -0.7 (0.07) | -0.7 (0.09)
  Change at Final Week (AM) | -0.6 (0.07) | -0.6 (0.08)
  Baseline (PM) | 1.7 (0.06) | 1.6 (0.07)
  Change at Week 1 (PM) | -0.3 (0.06) | -0.4 (0.07)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -0.4 (0.06) | -0.5 (0.07)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -0.6 (0.07) | -0.6 (0.08)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -0.7 (0.07) | -0.7 (0.09)
  Change at Final Week (PM) | -0.6 (0.07) | -0.6 (0.08)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.078, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.492, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.945, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.359, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.802, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.716, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.158, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.281, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.901, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.433, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.730, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.819, ANOVA

5. Secondary Outcome: Change From Baseline in AM and PM Chest Tightness Symptom Score
Description: Chest tightness is an asthma symptom assessed by participants using diary cards to record morning and evening chest tightness (recorded twice daily). Every morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her chest tightness for the time period since the last evaluation (or for the previous 12 hours for the first evaluation). The severity of chest tightness was rated on a 4-point scale (0=no symptom [best score] to 3=symptoms were hard to tolerate and interfered with daily life activity [worst score]). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 1.6 (0.07) | 1.6 (0.08)
  Change at Week 1 (AM) | -0.2 (0.06) | -0.4 (0.07)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -0.3 (0.08) | -0.4 (0.09)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -0.5 (0.07) | -0.7 (0.08)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -0.5 (0.07) | -0.7 (0.08)
  Change at Final Week (AM) | -0.4 (0.07) | -0.6 (0.08)
  Baseline (PM) | 1.6 (0.07) | 1.6 (0.08)
  Change at Week 1 (PM) | -0.3 (0.06) | -0.5 (0.07)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -0.4 (0.07) | -0.5 (0.08)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -0.6 (0.07) | -0.7 (0.08)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -0.6 (0.07) | -0.7 (0.08)
  Change at Final Week (PM) | -0.6 (0.06) | -0.6 (0.08)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.629, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.038, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.182, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.149, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.035, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.056, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.711, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.098, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.356, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.529, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.617, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.422, ANOVA

6. Secondary Outcome: Change From Baseline in Pulmonary Auscultation/Wheezing Assessment
Description: Wheezing was assessed by the investigator or designee based upon pulmonary auscultation (listening with a stethoscope) and reported in the case report form as present or absent. The count of wheezing presence (yes, no) at visits was summarized.
Time Frame: Baseline, Day 15 and Day 29
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Participants
  Present at Baseline | 11 | 9
  Absent at Baseline | 101 | 66
  Present on Day 15: number analyzed (Participants) | 102 | 72
  Present on Day 15 | 8 | 4
  Absent on Day 15: number analyzed (Participants) | 102 | 72
  Absent on Day 15 | 94 | 68
  Present on Day 29: number analyzed (Participants) | 108 | 74
  Present on Day 29 | 10 | 3
  Absent on Day 29: number analyzed (Participants) | 108 | 74
  Absent on Day 29 | 98 | 71
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Baseline; p = 0.532, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Day 15; p = 0.739, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Day 29; p = 0.227, Cochran-Mantel-Haenszel

7. Secondary Outcome: Change From Baseline in AM and PM Total Nasal Symptom Severity (TNSS)
Description: The Total Nasal Symptom Severity (TNSS) is the sum of severity scores for 4 nasal symptoms: nasal rhinorrhea, nasal stuffiness/congestion, sneezing, and nasal itching as assessed in the participant diaries. The severity of each nasal symptom was rated on a 4-point scale (0=no symptom [best score] to 3=symptoms were hard to tolerate and interfered with daily life activity [worst score]); minimum TNSS=0; maximum TNSS=12. A decrease in TNSS indicated an improvement in nasal symptoms. The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 8.4 (0.19) | 7.9 (0.23)
  Week 1 (AM) | -1.7 (0.21) | -0.9 (0.25)
  Week 2 (AM): number analyzed (Participants) | 109 | 75
  Week 2 (AM) | -2.3 (0.27) | -1.3 (0.30)
  Week 3 (AM): number analyzed (Participants) | 98 | 71
  Week 3 (AM) | -3.2 (0.29) | -1.8 (0.32)
  Week 4 (AM): number analyzed (Participants) | 98 | 69
  Week 4 (AM) | -3.5 (0.32) | -2.4 (0.37)
  Final Week (AM) | -3.1 (0.29) | -2.2 (0.35)
  Baseline (PM) | 8.2 (0.20) | 7.9 (0.23)
  Week 1 (PM) | -1.8 (0.22) | -1.5 (0.25)
  Week 2 (PM): number analyzed (Participants) | 110 | 75
  Week 2 (PM) | -2.6 (0.26) | -1.8 (0.30)
  Week 3 (PM): number analyzed (Participants) | 100 | 71
  Week 3 (PM) | -3.4 (0.28) | -2.4 (0.31)
  Week 4 (PM): number analyzed (Participants) | 98 | 69
  Week 4 (PM) | -3.6 (0.31) | -2.8 (0.36)
  Final Week (PM) | -3.3 (0.30) | -2.6 (0.35)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.104, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.022, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.012, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.001, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.033, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.047, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.269, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.308, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.050, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.014, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.100, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.139, ANOVA

8. Secondary Outcome: Change From Baseline in AM and PM Rhinorrhea Symptom Score
Description: Rhinorrhea is a symptom of seasonal allergic rhinitis (SAR) assessed by participants using diary cards to record morning and evening rhinorrhea (recorded twice daily). Every morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her rhinorrhea for the time period since the last evaluation (or for the previous 12 hours for the first evaluation). Rhinorrhea was assessed on a 4-point scale (0=no symptom [best score] to 3=symptoms were hard to tolerate and interfered with daily life activity [worst score]). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 2.2 (0.06) | 2.1 (0.07)
  Change at Week 1 (AM) | -0.3 (0.06) | -0.2 (0.07)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -0.5 (0.08) | -0.3 (0.09)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -0.7 (0.09) | -0.4 (0.10)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -0.9 (0.09) | -0.5 (0.11)
  Change at Final Week (AM) | -0.8 (0.09) | -0.5 (0.10)
  Baseline (PM) | 2.1 (0.06) | 2.0 (0.07)
  Change at Week 1 (PM) | -0.4 (0.06) | -0.3 (0.07)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -0.5 (0.07) | -0.4 (0.08)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -0.8 (0.08) | -0.5 (0.09)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -0.9 (0.09) | -0.6 (0.10)
  Change at Final Week (PM) | -0.8 (0.08) | -0.5 (0.10)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.136, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.126, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.107, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.006, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.030, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.037, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.146, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.426, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.259, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.026, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.022, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.043, ANOVA

9. Secondary Outcome: Change From Baseline in AM and PM Nasal Itching Symptom Score
Description: Nasal itching is a symptom of SAR assessed by participants using diary cards to record morning and evening nasal itching (recorded twice daily). Every morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her nasal itching for the time period since the last evaluation (or for the previous 12 hours for the first evaluation). It was assessed on a 4-point scale (0=no symptom [best score] to 3=symptoms were hard to tolerate and interfered with daily life activity [worst score]). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 2.0 (0.07) | 1.9 (0.08)
  Change at Week 1 (AM) | -0.4 (0.07) | -0.2 (0.08)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -0.6 (0.08) | -0.3 (0.09)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -0.9 (0.08) | -0.5 (0.09)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -0.9 (0.09) | -0.6 (0.11)
  Change at Final Week (AM) | -0.8 (0.09) | -0.5 (0.10)
  Baseline (PM) | 1.7 (0.07) | 1.5 (0.08)
  Change at Week 1 (PM) | -0.4 (0.06) | -0.3 (0.07)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -0.7 (0.07) | -0.4 (0.09)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -0.9 (0.08) | -0.6 (0.09)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -0.9 (0.09) | -0.7 (0.11)
  Change at Final Week (PM) | -0.8 (0.09) | -0.6 (0.10)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.181, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.014, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.004, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.002, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.027, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.069, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.373, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.148, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.009, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.016, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.113, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.173, ANOVA

10. Secondary Outcome: Change From Baseline in AM and PM Nasal Sneezing Symptom Score
Description: Nasal sneezing is a symptom of SAR assessed by participants using diary cards to record morning and evening nasal sneezing (recorded twice daily). Every morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her nasal sneezing for the time period since the last evaluation (or for the previous 12 hours for the first evaluation). It was assessed on a 4-point scale (0=no symptom [best score] to 3=symptoms a were hard to tolerate and interfered with daily life activity [worst score]). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 1.8 (0.07) | 1.7 (0.08)
  Change at Week 1 (AM) | -0.5 (0.07) | -0.2 (0.08)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -0.6 (0.08) | -0.6 (0.09)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -0.9 (0.08) | -0.4 (0.09)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -0.9 (0.09) | -0.6 (0.10)
  Change at Final Week (AM) | -0.8 (0.08) | -0.6 (0.10)
  Baseline (PM) | 1.9 (0.06) | 1.8 (0.08)
  Change at Week 1 (PM) | -0.5 (0.07) | -0.4 (0.08)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -0.7 (0.08) | -0.5 (0.09)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -0.9 (0.08) | -0.6 (0.09)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -0.9 (0.09) | -0.7 (0.11)
  Change at Final Week (PM) | -0.9 (0.08) | -0.7 (0.10)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.089, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.014, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.004, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.001, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.041, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.036, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.170, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.237, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.019, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.018, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.149, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.231, ANOVA

11. Secondary Outcome: Change From Baseline in AM and PM Nasal Congestion Symptom Score
Description: Nasal congestion is a symptom of SAR assessed by participants using diary cards to record morning and evening nasal congestion (recorded twice daily). Every morning prior to dosing and each evening approximately 12 hours later, the participant evaluated his/her nasal congestion for the time period since the last evaluation (or for the previous 12 hours for the first evaluation). It was assessed on a 4-point scale (0=no symptom [best score] to 3=symptoms were hard to tolerate and interfered with daily life activity [worst score]). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline (AM) | 2.3 (0.05) | 2.3 (0.06)
  Change at Week 1 (AM) | -0.4 (0.06) | -0.3 (0.07)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | -0.5 (0.07) | -0.4 (0.08)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | -0.7 (0.08) | -0.5 (0.09)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | -0.8 (0.10) | -0.7 (0.11)
  Change at Final Week (AM) | -0.8 (0.08) | -0.6 (0.10)
  Baseline (PM) | 2.2 (0.05) | 2.2 (0.06)
  Change at Week 1 (PM) | -0.4 (0.07) | -0.4 (0.08)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | -0.6 (0.08) | -0.5 (0.09)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | -0.8 (0.08) | -0.6 (0.09)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | -0.9 (0.09) | -0.8 (0.11)
  Change at Final Week (PM) | -0.8 (0.09) | -0.7 (0.10)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.745, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.250, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Week 2 (AM); p = 0.202, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Week 3 (AM); p = 0.104, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Week 4 (AM); p = 0.348, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Final Week (AM); p = 0.355, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Baseline (PM); p = 0.851, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Week 1 (PM); p = 0.993, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Week 2 (PM); p = 0.476, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Week 3 (PM); p = 0.149, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Week 4 (PM); p = 0.616, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Test type: Superiority or Other — Change at Final Week (PM); p = 0.527, ANOVA

12. Secondary Outcome: Change From Baseline in AM and PM Peak Expiratory Flow Rate (PEFR)
Description: Participants used a peak flow meter to measure the rate of air forcibly expelled from the lungs. They performed triplicate PEFR measurements in the morning prior to taking their study medication and again in the evening, and documented the highest of the three values in their diaries. A day with worsening asthma was any day during which a decrease from baseline in morning (AM) PEFR of more than 25% occurred. The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Liters/min
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Liters/min
  Baseline (AM) | 382.5 (8.35) | 362.3 (9.97)
  Change at Week 1 (AM) | 0.9 (2.83) | 1.0 (3.34)
  Change at Week 2 (AM): number analyzed (Participants) | 109 | 75
  Change at Week 2 (AM) | 4.3 (3.28) | 4.1 (3.74)
  Change at Week 3 (AM): number analyzed (Participants) | 98 | 71
  Change at Week 3 (AM) | 7.7 (3.34) | 1.0 (3.73)
  Change at Week 4 (AM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (AM) | 7.8 (3.79) | 3.3 (4.35)
  Change at Final Week (AM) | 5.7 (3.37) | 4.6 (3.97)
  Baseline (PM) | 394.4 (8.18) | 373.4 (9.77)
  Change at Week 1 (PM) | 0.5 (2.67) | 4.3 (3.15)
  Change at Week 2 (PM): number analyzed (Participants) | 110 | 75
  Change at Week 2 (PM) | 4.9 (3.43) | 7.0 (3.96)
  Change at Week 3 (PM): number analyzed (Participants) | 100 | 71
  Change at Week 3 (PM) | 5.8 (3.70) | 8.7 (4.19)
  Change at Week 4 (PM): number analyzed (Participants) | 98 | 69
  Change at Week 4 (PM) | 6.9 (4.08) | 10.3 (4.69)
  Change at Final Week (PM) | 5.6 (3.58) | 10.1 (4.22)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline (AM); Test type: Superiority or Other; p = 0.116, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1 (AM); Test type: Superiority or Other; p = 0.994, ANOVA
Statistical Analysis 3: Comparison: Mometasone; Change at Week 2 (AM); Test type: Superiority or Other; p = 0.961, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3 (AM); Test type: Superiority or Other; p = 0.183, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4 (AM); Test type: Superiority or Other; p = 0.440, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week (AM); Test type: Superiority or Other; p = 0.838, ANOVA
Statistical Analysis 7: Comparison: Mometasone vs Placebo; Baseline (PM); Test type: Superiority or Other; p = 0.096, ANOVA
Statistical Analysis 8: Comparison: Mometasone vs Placebo; Change at Week 1 (PM); Test type: Superiority or Other; p = 0.362, ANOVA
Statistical Analysis 9: Comparison: Mometasone vs Placebo; Change at Week 2 (PM); Test type: Superiority or Other; p = 0.693, ANOVA
Statistical Analysis 10: Comparison: Mometasone vs Placebo; Change at Week 3 (PM); Test type: Superiority or Other; p = 0.603, ANOVA
Statistical Analysis 11: Comparison: Mometasone vs Placebo; Change at Week 4 (PM); Test type: Superiority or Other; p = 0.579, ANOVA
Statistical Analysis 12: Comparison: Mometasone vs Placebo; Change at Final Week (PM); Test type: Superiority or Other; p = 0.413, ANOVA

13. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1)
Description: Measured by the investigator (or a designated assistant) using a spirometer, FEV1 is the volume of air forcibly expelled from the lungs in one second.
Time Frame: Baseline, Day 15 and Day 29
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Liters
  Baseline | 2.98 (0.06) | 3.00 (0.07)
  Change at Day 15: number analyzed (Participants) | 103 | 72
  Change at Day 15 | 0.05 (0.03) | 0.07 (0.04)
  Change at Day 29: number analyzed (Participants) | 108 | 74
  Change at Day 29 | 0.04 (0.04) | 0.02 (0.04)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline; Test type: Superiority or Other; p = 0.823, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Day 15; Test type: Superiority or Other; p = 0.744, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Day 29; Test type: Superiority or Other; p = 0.675, ANOVA

14. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: Measured by the investigator (or a designated assistant) using a spirometer, FVC is the total volume of air forcibly expelled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Day 15 and Day 29
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Liters
  Baseline | 3.75 (0.08) | 3.80 (0.10)
  Change at Day 15: number analyzed (Participants) | 103 | 72
  Change at Day 15 | 0.02 (0.03) | 0.00 (0.04)
  Change at Day 29: number analyzed (Participants) | 108 | 74
  Change at Day 29 | -0.00 (0.04) | 0.00 (0.04)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline; Test type: Superiority or Other; p = 0.693, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Day 15; Test type: Superiority or Other; p = 0.818, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Day 29; Test type: Superiority or Other; p = 0.915, ANOVA

15. Secondary Outcome: Change From Baseline in Forced Expiratory Flow (FEF) Between 25% and 75% of the Vital Capacity (FEF25%-75%)
Description: Measured by the investigator (or a designated assistant) using a spirometer, FEF25%-75% is the average forcibly expelled air flow rate, measured between 75% and 25% of FVC.
Time Frame: Baseline, Day 15 and Day 29
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Liters/sec
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Liters/sec
  Baseline | 2.98 (0.06) | 3.00 (0.07)
  Change at Day 15: number analyzed (Participants) | 103 | 72
  Change at Day 15 | 0.12 (0.06) | 0.00 (0.07)
  Change at Day 29: number analyzed (Participants) | 108 | 74
  Change at Day 29 | 0.15 (0.06) | 0.03 (0.07)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline; Test type: Superiority or Other; p = 0.823, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Day 15; Test type: Superiority or Other; p = 0.202, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Day 29; Test type: Superiority or Other; p = 0.199, ANOVA

16. Secondary Outcome: Change From Baseline in the Weekly Average Number of Puffs of Albuterol/Salbutamol Used
Description: Once daily, participants recorded in their diaries the total number of puffs of albuterol/salbutamol used in each 24-hour period. The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Number of puffs
  Baseline | 2.4 (0.18) | 2.1 (0.21)
  Change at Week 1 | -0.4 (0.14) | -0.5 (0.17)
  Change at Week 2: number analyzed (Participants) | 111 | 75
  Change at Week 2 | -0.6 (0.16) | -0.5 (0.18)
  Change at Week 3: number analyzed (Participants) | 101 | 72
  Change at Week 3 | -0.8 (0.15) | -0.5 (0.17)
  Change at Week 4: number analyzed (Participants) | 98 | 69
  Change at Week 4 | -0.7 (0.17) | -0.6 (0.19)
  Change at Final Week | -0.7 (0.16) | -0.6 (0.19)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline; Test type: Superiority or Other; p = 0.375, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1; Test type: Superiority or Other; p = 0.710, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2; Test type: Superiority or Other; p = 0.597, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3; Test type: Superiority or Other; p = 0.242, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4; Test type: Superiority or Other; p = 0.696, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week; Test type: Superiority or Other; p = 0.670, ANOVA

17. Secondary Outcome: Change From Baseline in Weekly Average Nighttime Awakenings Due to Asthma
Description: Participants recorded the number of times during the night they awakened due to asthma. The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Awakenings
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Awakenings
  Baseline | 0.6 (0.08) | 0.6 (0.09)
  Change at Week 1 | -0.1 (0.05) | -0.2 (0.06)
  Change at Week 2: number analyzed (Participants) | 111 | 74
  Change at Week 2 | -0.1 (0.06) | -0.2 (0.07)
  Change at Week 3: number analyzed (Participants) | 103 | 74
  Change at Week 3 | -0.3 (0.07) | -0.3 (0.08)
  Change at Week 4: number analyzed (Participants) | 98 | 68
  Change at Week 4 | -0.2 (0.07) | -0.3 (0.08)
  Change at Final Week | -0.2 (0.06) | -0.3 (0.07)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline; Test type: Superiority or Other; p = 0.865, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1; Test type: Superiority or Other; p = 0.025, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2; Test type: Superiority or Other; p = 0.288, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3; Test type: Superiority or Other; p = 0.790, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4; Test type: Superiority or Other; p = 0.211, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week; Test type: Superiority or Other; p = 0.136, ANOVA

18. Secondary Outcome: Change From Baseline in Weekly Average Interference With Sleep
Description: Interference with sleep was rated once each morning using a 4-point scale ranging from 0 (none) to 3 (substantially interferes with sleep). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline | 1.3 (0.07) | 1.2 (0.09)
  Change at Week 1 | -0.2 (0.05) | -0.2 (0.06)
  Change at Week 2: number analyzed (Participants) | 111 | 75
  Change at Week 2 | -0.4 (0.07) | -0.3 (0.08)
  Change at Week 3: number analyzed (Participants) | 103 | 75
  Change at Week 3 | -0.5 (0.06) | -0.4 (0.07)
  Change at Week 4: number analyzed (Participants) | 98 | 69
  Change at Week 4 | -0.5 (0.07) | -0.5 (0.08)
  Change at Final Week | -0.4 (0.07) | -0.4 (0.08)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline; Test type: Superiority or Other; p = 0.667, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1; Test type: Superiority or Other; p = 0.656, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2; Test type: Superiority or Other; p = 0.458, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3; Test type: Superiority or Other; p = 0.220, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4; Test type: Superiority or Other; p = 0.775, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week; Test type: Superiority or Other; p = 0.994, ANOVA

19. Secondary Outcome: Change From Baseline in Weekly Average Interference With Daily Activities
Description: Interference with daily activities was rated once each evening using a 4-point scale ranging from 0 (none) to 3 (substantially interfered with activities or not able to perform the activities at all). The Final Week was the final 7 days post Day 1 (e. g., if Day 20 was the day of last dose of study medication, then the AM assessment at Final Week was calculated from Day 14 to Day 20, and the PM assessment at Final Week was calculated from Day 13 to Day 19).
Time Frame: Baseline up to Week 4
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Baseline | 1.5 (0.06) | 1.4 (0.08)
  Change at Week 1: number analyzed (Participants) | 111 | 75
  Change at Week 1 | -0.3 (0.05) | -0.4 (0.06)
  Change at Week 2: number analyzed (Participants) | 107 | 75
  Change at Week 2 | -0.4 (0.06) | -0.3 (0.07)
  Change at Week 3: number analyzed (Participants) | 98 | 70
  Change at Week 3 | -0.6 (0.07) | -0.4 (0.07)
  Change at Week 4: number analyzed (Participants) | 98 | 67
  Change at Week 4 | -0.6 (0.08) | -0.5 (0.09)
  Change at Final Week | -0.5 (0.07) | -0.5 (0.08)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Baseline; Test type: Superiority or Other; p = 0.363, ANOVA
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Change at Week 1; Test type: Superiority or Other; p = 0.262, ANOVA
Statistical Analysis 3: Comparison: Mometasone vs Placebo; Change at Week 2; Test type: Superiority or Other; p = 0.386, ANOVA
Statistical Analysis 4: Comparison: Mometasone vs Placebo; Change at Week 3; Test type: Superiority or Other; p = 0.167, ANOVA
Statistical Analysis 5: Comparison: Mometasone vs Placebo; Change at Week 4; Test type: Superiority or Other; p = 0.505, ANOVA
Statistical Analysis 6: Comparison: Mometasone vs Placebo; Change at Final Week; Test type: Superiority or Other; p = 0.725, ANOVA

20. Secondary Outcome: Therapeutic Response to Asthma Symptoms
Description: On Day 15 and Day 29, the investigator or designee and participant jointly assessed the participant's response to study intervention by comparing the current level of asthma symptoms with those noted on Day 1. Therapeutic response for asthma symptoms was based on a 5-point scale ranging from 1 (Complete Relief) to 5 (No Relief).
Time Frame: Day 15 and Day 29
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  Asthma: Day 15: number analyzed (Participants) | 103 | 71
  Asthma: Day 15 | 3.4 (1.13) | 3.4 (1.05)
  Asthma: Day 29: number analyzed (Participants) | 109 | 74
  Asthma: Day 29 | 3.2 (1.26) | 3.5 (1.14)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Asthma Symptoms: Day 15; Test type: Superiority or Other; p = 0.954, Cochran-Mantel-Haenszel; Stratified by center
Statistical Analysis 2: Comparison: Mometasone vs Placebo; Asthma Symptoms: Day 29; Test type: Superiority or Other; p = 0.295, Cochran-Mantel-Haenszel; Stratified by center

21. Secondary Outcome: Therapeutic Response to SAR Nasal Symptoms
Description: On Day 15 and Day 29, the investigator or designee and participant jointly assessed the participant's response to study intervention by comparing the current level of SAR symptoms with those noted on Day 1. Therapeutic response for SAR symptoms was based on a 5-point scale ranging from 1 (Complete Relief) to 5 (No Relief).
Time Frame: Day 15 and Day 29
Population: All randomized participants who had at least one post-baseline assessment at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 112 | 75
Score on a scale
  SAR Nasal: Day 15: number analyzed (Participants) | 103 | 71
  SAR Nasal: Day 15 | 3.2 (1.11) | 3.4 (1.01)
  SAR Nasal: Day 29: number analyzed (Participants) | 109 | 74
  SAR Nasal: Day 29 | 3.0 (1.13) | 3.4 (1.04)
Statistical Analysis 1: Comparison: Mometasone vs Placebo; SAR Nasal Symptoms: Day 15; Test type: Superiority or Other; p = 0.268, Cochran-Mantel-Haenszel; Stratified by center
Statistical Analysis 2: Comparison: Mometasone vs Placebo; SAR Nasal Symptoms: Day 29; Test type: Superiority or Other; p = 0.154, Cochran-Mantel-Haenszel; Stratified by center

ADVERSE EVENTS:
Time Frame: Up to 59 days
Description: An AE is any physical or clinical change or disease the participant experiences at any time during the course of the study, whether or not considered related to the use of the study drug. The population analyzed is all randomized participants who receive at least one dose of treatment.
Arm/Group | Mometasone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/113 | 1/75
Other Adverse Events (participants affected / at risk) | 4/113 | 4/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone (N=113) | Placebo (N=75)
Fracture, bone (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone (N=113) | Placebo (N=75)
Headache (General disorders) | 4 (5) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Manuscript(s) and abstract(s) were prepared through cooperation between the sponsor and the study investigator(s). The principal investigator (PI) had the right to publish or publicly present the Study results. The PI agreed to provide thirty (30) days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of abstracts or manuscripts for publication. The sponsor had the right to review and comment on any publication.